CLINICAL TRIAL: NCT00041496
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Group Study of the Safety and Efficacy of SB 207266 in Patients With Symptomatic Persistent Atrial Fibrillation (AF)
Brief Title: Prevention Of Recurrence Of Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 207266082
Record Dates: First submitted 2002-07-09; First posted 2002-07-12 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Fibrillation, Atrial
Keywords: symptomatic atrial fibrillation; persistent atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — SB 207266

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental): Patients with Symptomatic Persistent Atrial Fibrillation (AF) will be randomized with either SB207266 or placebo
  Interventions: Drug: SB-207266
- Arm 2 (Placebo Comparator): Patients with Symptomatic Persistent Atrial Fibrillation (AF) will be randomized with either SB207266 or Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SB-207266 — White, oval, biconvex tablets containing either 10mg, 25mg or 40mg
  Arms: Arm 1
Other: Placebo — Placebo to match SB-207266
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine whether the study drug is effective in preventing the recurrence of atrial fibrillation (an abnormal heart rhythm).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic persistent atrial fibrillation requiring DC cardioversion.
* Duration of AF >48 hrs. <6 months

Exclusion Criteria:

* Concomitant Class I and/or III anti-arrhythmic drugs.
* Amiodarone treatment within 3 months of the study.
* Other inclusion or exclusion criteria to be determined by the physician and study sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2001-11; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Time-to-first symptomatic AF (atrial fibrillation) | Up to 26 Weeks

SECONDARY OUTCOMES:
Time to first symptomatic or detected asymptomatic AF; spontaneous reversion to sinus rhythm prior to cardioversion | Up to 26 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline